CLINICAL TRIAL: NCT06535594
Title: The Potential Efficacy Of Laser Acupuncture Combined With Physiotherapy In Managing Pain And Improve The Elbow Active Range Of Motions Improve The Elbow Active Range Of Motion In 30 Tennis Elbow Syndrome Patients: A Pre - Post Trial
Brief Title: Efficacy Of Laser Acupuncture Combined With Physiotherapy In Tennis Elbow Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Do Thanh Sang, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 271/HDDD-DHYD
Record Dates: First submitted 2024-07-27; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser acupuncture + Physical therapy (Experimental): Laser acupuncture five times a week for a total of four weeks (20 sessions). Physical therapy three times a day, five times a week for a total of four weeks.
  Interventions: Other: Laser acupuncture; Other: Physical therapy

INTERVENTIONS:
Other: Laser acupuncture — Laser acupuncture therapy will be performed five times a week for 4 weeks using laser beam. The acupoints on the ear that will be treated with laser acupuncture therapy are Zhouliao (LI12), Chize (LU5), Quchi (LI11), Shousanli (LI10) and Ashi.
Other: Physical therapy — Physical therapy method involved six elbow joint exercises. Patients performed the six exercises sequentially under guidance, each exercise performed five times, three times a day, gradually increasing weight until the movement was effective but below the pain threshold.

SUMMARY:
Tennis Elbow (TE) syndrome affects 1 to 3% of adults annually. The burden of TE syndrome continues to increase annually due to repeated microtrauma to the forearm extensor tendon. Treatment mainly includes anti-inflammatory pain medications, physical therapy, shockwave therapy, Laser acupuncture therapy, topical nitrates, elbow braces, and corticosteroid injections. Surgery is considered for cases where conservative treatment fails, including open and arthroscopic surgery.

Laser acupuncture (LA) is a new acupuncture technique using Laser beams to stimulate acupuncture points, offering a less invasive alternative to traditional needles and demonstrating therapeutic effectiveness. Recent Studies have shown that LA significantly improves pain in TE patients. Additionally, combining physical therapy for functional rehabilitation in treating TE syndrome plays an essential role in alleviating pain and restoring elbow joint function, preventing long-term stiffness. In practice, many hospitals apply a combination of LA and physical therapy to treat TE with considerable effectiveness, though it has not been thoroughly evidence-based.

Given the limitations in evaluating treatment effectiveness and the lack of published research discussing the analgesic effects of LA for TE syndrome, as well as to enhance the effectiveness of combining TCM and modern medicine, the investigators conducted the study Pain Reduction and Range of Motion Improvement of LA Combined with Physical Therapy in Patients with TE syndrome.

DETAILED DESCRIPTION:
Patients with Tennis Elbow syndrome who have main symptoms such as pain and tenderness at the lateral epicondyle or radial head will be registered for this study. They will be treated with a combination of Laser acupuncture and physical therapy.

The intervention period is four weeks. Laser acupuncture and physical therapy will be performed five times a week.

Data on the Visual Analog Scale (VAS), Active range of motion of the elbow joint, and side effects of Laser acupuncture and physical therapy will be recorded before the study and weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 19 and 65 years with Tennis Elbow in one arm and pain persisting for at least 4 weeks.
* Individuals with tenderness limited to the elbow joint and surrounding area.
* Individuals reporting pain under resisted extension of the middle finger and wrist.
* Individuals with an average pain score of 4 or more (0-10) on the Visual Analogue Scale (VAS) in the week prior to the screening visit.
* Individuals who volunteered to participate in the study and signed a consent form.
* Experiencing elbow pain for more than four weeks.

Exclusion Criteria:

* Patients with previous elbow surgery, systemic diseases affecting joint mobility, or those who received any form of treatment for TE in the last three months.
* Patients requiring elbow joint replacement surgery.
* Patients with psychiatric disorders.
* Patients with elbow-related conditions other than TE: elbow trauma, elbow tuberculosis, cancer.
* Patients with unexplained skin abnormalities around the elbow joint, currently using immunosuppressive drugs, or on prolonged corticosteroid treatment.
* Patients with an acute illness requiring prior intervention.
* Individuals with a history of trauma, ligament damage, fracture, tumor, or surgery of the elbow joint.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The change of the Visual Analog Scale (VAS) | Assessments were conducted before intervention and after each intervention week throughout the four weeks (Week 0, Week 1, Week 2, Week 3, Week 4)
  Symptom scores will be assessed based on a visual analogue scale (VAS). It usually consists of a 10 cm line anchored at each end by descriptors. Patients will be classified into 1 of 4 groups (no pain (0 cm), mild pain (1-3 cm), moderate pain (4-7 cm), severe pain (8-10 cm)).

SECONDARY OUTCOMES:
Proportion of intervention-related adverse events | Up to four weeks
  While laser acupuncture is generally considered safe, some patients may experience minor side effects at the application site. These can include skin redness or burns. Rarely, more serious complications like dizziness, headaches, and fatigue may occur. The study will closely monitor and document any unexpected adverse events associated with the procedure.
The change of active range of motion of the elbow joint | Assessments were conducted before intervention and after each intervention week throughout the four weeks (Week 0, Week 1, Week 2, Week 3, Week 4)
  Active range of motion of the elbow joint measured using a goniometer.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quah-Smith I, Williams MA, Lundeberg T, Suo C, Sachdev P. Differential brain effects of laser and needle acupuncture at LR8 using functional MRI. Acupunct Med. 2013 Sep;31(3):282-9. doi: 10.1136/acupmed-2012-010297. Epub 2013 Aug 6. PMID 23920052
- [Background] Haker E, Lundeberg T. Laser treatment applied to acupuncture points in lateral humeral epicondylalgia. A double-blind study. Pain. 1990 Nov;43(2):243-247. doi: 10.1016/0304-3959(90)91078-W. PMID 2087335
- [Background] Yoon SY, Kim YW, Shin IS, Kang S, Moon HI, Lee SC. The Beneficial Effects of Eccentric Exercise in the Management of Lateral Elbow Tendinopathy: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 1;10(17):3968. doi: 10.3390/jcm10173968. PMID 34501416
- [Background] Dingemanse R, Randsdorp M, Koes BW, Huisstede BM. Evidence for the effectiveness of electrophysical modalities for treatment of medial and lateral epicondylitis: a systematic review. Br J Sports Med. 2014 Jun;48(12):957-65. doi: 10.1136/bjsports-2012-091513. Epub 2013 Jan 18. PMID 23335238
- [Background] Zhou Y, Guo Y, Zhou R, Wu P, Liang F, Yang Z. Effectiveness of Acupuncture for Lateral Epicondylitis: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pain Res Manag. 2020 Mar 20;2020:8506591. doi: 10.1155/2020/8506591. eCollection 2020. PMID 32318130
- [Background] Adly AS, Adly AS, Adly MS. Effects of laser acupuncture tele-therapy for rheumatoid arthritis elderly patients. Lasers Med Sci. 2022 Feb;37(1):499-504. doi: 10.1007/s10103-021-03287-0. Epub 2021 Mar 19. PMID 33738615
- [Background] Bisset L, Beller E, Jull G, Brooks P, Darnell R, Vicenzino B. Mobilisation with movement and exercise, corticosteroid injection, or wait and see for tennis elbow: randomised trial. BMJ. 2006 Nov 4;333(7575):939. doi: 10.1136/bmj.38961.584653.AE. Epub 2006 Sep 29. PMID 17012266
- [Background] Yi R, Bratchenko WW, Tan V. Deep Friction Massage Versus Steroid Injection in the Treatment of Lateral Epicondylitis. Hand (N Y). 2018 Jan;13(1):56-59. doi: 10.1177/1558944717692088. Epub 2017 Feb 1. PMID 28719982
- [Background] Ciccotti MC, Schwartz MA, Ciccotti MG. Diagnosis and treatment of medial epicondylitis of the elbow. Clin Sports Med. 2004 Oct;23(4):693-705, xi. doi: 10.1016/j.csm.2004.04.011. PMID 15474230
- [Background] Degen RM, Conti MS, Camp CL, Altchek DW, Dines JS, Werner BC. Epidemiology and Disease Burden of Lateral Epicondylitis in the USA: Analysis of 85,318 Patients. HSS J. 2018 Feb;14(1):9-14. doi: 10.1007/s11420-017-9559-3. Epub 2017 Jun 5. PMID 29398988
- [Background] Duncan J, Duncan R, Bansal S, Davenport D, Hacker A. Lateral epicondylitis: the condition and current management strategies. Br J Hosp Med (Lond). 2019 Nov 2;80(11):647-651. doi: 10.12968/hmed.2019.80.11.647. PMID 31707890